CLINICAL TRIAL: NCT03442621
Title: A Phase 1, Open-label, Single-dose, Randomized, Crossover Study in Healthy Subjects of the Effects of Co-administration With Food on Exposure, and to Determine the Within-subject Variability in Exposure, to Relacorilant and Its Metabolites
Brief Title: Relacorilant Food Effect Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CORT125134-123
Record Dates: First submitted 2018-01-23; First posted 2018-02-22 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-02

CONDITIONS: Healthy; Food-drug Interaction
MeSH Terms: interventions — relacorilant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Relacorilant Fasted (Experimental): Relacorilant Fasted
  Interventions: Drug: Relacorilant Fasted
- Relacorilant with a high fat breakfast (Experimental): Relacorilant with a high fat breakfast
  Interventions: Drug: Relacorilant with a high fat breakfast
- Relacorilant with a moderate breakfast (Experimental): Relacorilant with a moderate breakfast
  Interventions: Drug: Relacorilant with a moderate breakfast

INTERVENTIONS:
Drug: Relacorilant Fasted — Relacorilant, presented as 7 x 50-mg white, hard gelatin capsules for oral administration, given following a 10.5 h fast
  Other Names: Relacorilant; CORT125134
  Arms: Relacorilant Fasted
Drug: Relacorilant with a high fat breakfast — Relacorilant presented as 7 x 50-mg white, hard gelatin capsules for oral administration, given following a 10 h fast and 0.5 h after the start of a high fat breakfast
  Other Names: Relacorilant; CORT125134
  Arms: Relacorilant with a high fat breakfast
Drug: Relacorilant with a moderate breakfast — Relacorilant, presented as 7 x 50-mg white, hard gelatin capsules for oral administration, given following a 10 h fast and 0.5 h after the start of a moderate breakfast
  Other Names: Relacorilant; CORT125134
  Arms: Relacorilant with a moderate breakfast

SUMMARY:
This is an open-label, randomized, single-dose, 3-period crossover, Williams' design, food-interaction (fasted and fed arms) study conducted in healthy subjects.

DETAILED DESCRIPTION:
This food-interaction study will be conducted in healthy subjects. Each subject will have a screening visit (within the 21 days prior to the first study drug administration to confirm eligibility), 3 single-dose treatment periods separated by a 7- to 14- day washout between doses, and an outpatient end-of-study follow-up visit 14 +/- 2 days after the last dose of study medication. During each treatment period, subjects will receive a single 350-mg relacorilant dose. Based on randomization to 1 of 6 sequences, each subject will receive the relacorilant dose once after a 10.5 hour fast; once 30 minutes after the start of a high-fat meal; and once 30 minutes after the start of a moderate meal.

During the first treatment period only, regardless of randomized sequence, subjects will report to the clinical research unit on the morning of Day -1 for baseline laboratory assessments and to collect samples for assay of messenger ribonucleic acid (mRNA) expression of glucocorticoid-modulated genes to explore the normal range over the day in healthy subjects. For the subsequent 2 treatment periods, subjects will report to the CRU on the evening of Day -1.

Blood samples for assay of plasma concentration of relacorilant and its main metabolites will be collected pre-dose and at 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, and 96 hours post-dose. Subjects and will remain in the clinic until after the 24-hour blood samples are collected and then be discharged and scheduled to return for the later samples.

Additional samples will be collected for possible future pharmacogenomic analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the purpose and risks of the study; willing and able to adhere to scheduled visits, treatment plans, laboratory tests, and other study evaluations and procedures.
2. Give written informed consent.
3. Be males or nonpregnant, nonlactating females judged to be in good health, based on the results of medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory findings.
4. Have a body mass index (BMI) between 18 and 32 kg/m2, inclusive, and a body weight more than 50 kg (110 pounds).
5. Be a nonsmoker. Use of nicotine or nicotine-containing products must be discontinued at least 90 days prior to the first dose of study drug.
6. Be willing to comply with study restrictions
7. Have suitable veins for multiple venipuncture/cannulation.
8. Female subjects must be either of nonchildbearing potential (ie, postmenopausal or permanently sterilized) or use highly effective contraception with low user-dependency.

   * The only acceptable method of highly effective contraception with low user-dependency is an intrauterine device (IUD). Use of hormonal contraception (by any route, including intrauterine hormone releasing systems) or hormone replacement therapy is NOT acceptable.

Exclusion Criteria:

1. Be an employee or immediate family member of the Clinical Research Unit or Corcept.
2. Have been previously enrolled in any study of relacorilant.
3. Have multiple drug allergies, or be allergic to any of the components of relacorilant.
4. Have a condition that could be aggravated by glucocorticoid blockade (eg, asthma, any chronic inflammatory condition).
5. Have a history of gastric bypass surgery.
6. Have a history of malabsorption syndrome or previous gastrointestinal surgery, with the exception of appendectomy and cholecystectomy, which could affect drug absorption or metabolism.
7. Current alcohol or substance abuse.
8. In the 2 calendar months before first study drug administration, have donated/lost blood or plasma in excess of 400 mL.
9. In the 30 days before first study drug administration, have participated in another clinical trial of a new chemical entity or a prescription medicine.
10. Have a positive test for alcohol or drugs of abuse at screening or first admission.
11. Have a positive test for exogenous glucocorticoids at screening.
12. Have clinically relevant abnormal findings on vital signs, physical examination, laboratory screening tests, or 12-lead ECG, at screening and/or before first study drug administration, including but not limited to**:

    1. QT interval corrected for heart rate (QTc) using Fridericia's equation (QTcF) >450 ms (from mean of 3 supine ECGs, performed at least 2 minutes apart)
    2. Stage 2 or higher hypertension (supine/semi-recumbent systolic blood pressure [SBP] >160 mmHg, diastolic blood pressure [DBP] >100 mmHg; based on mean of duplicate values recorded at least 2 minutes apart)
    3. Stage 1 hypertension (supine/semi-recumbent SBP 140-160 mmHg, DBP 90-100 mmHg; based on mean of duplicate values recorded at least 2 minutes apart) associated with indication for treatment ie, evidence of end-organ damage, diabetes, or a 10-year cardiovascular risk, estimated using a standard calculator, (eg, QRISK2-2016) greater than 20%
    4. Glomerular filtration rate, estimated using the chronic kidney disease epidemiology (collaboration) (CKD-EPI) method (eGFR; Levey 2009) <60 mL/minute/1.73 m2
    5. Hypokalemia (potassium below lower limit of normal)
    6. Alanine aminotransferase (ALT), aspartate amino transferase (AST), and/or gamma- glutamyltransferase (GGT) >1.5 times the upper limit of normal (ULN)
    7. Seropositive for hepatitis B, hepatitis C, or human immunodeficiency (HIV) viruses **For purposes of qualifying any given subject for study participation, out-of-range values may be repeated once.
13. Have any medical or social reasons for not participating in the study raised by their primary care physician.
14. Have any other condition that might increase the risk to the individual or decrease the chance of obtaining satisfactory data, as assessed by the Investigator.
15. Taken any prohibited prior medication within protocol designated timeframes, such as or including any glucocorticoid, strong inducers, inhibitors or substrates of CYP enzymes involved in drug-drug-interactions, hormonal contraception or hormone replacement therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-03-09 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve up to the last quantifiable sample (AUC0-tz) | predose to 96 hrs postdose
  Ratio of population geometric means (GMR) for Test 1 (standard high fat breakfast) and Reference (fasted) and for Test 2 (standard moderate breakfast) and Reference for relacorilant areas under plasma concentration-time curve up to the last quantifiable sample (AUC0-tz)

SECONDARY OUTCOMES:
Area under plasma concentration-time curve extrapolated to infinity (AUCinf) | predose to 96 hrs postdose
  Ratio of population geometric means (GMR) for Test 1 (standard high fat breakfast) and Reference (fasted) and for Test 2 (standard moderate breakfast) and Reference for relacorilant areas under plasma concentration-time curve extrapolated to infinity (AUCinf)
Maximum plasma concentration (Cmax) | predose to 96 hrs postdose
  Ratio of population geometric means (GMR) for Test 1 (standard high fat breakfast) and Reference (fasted) and for Test 2 (standard moderate breakfast) and Reference for relacorilant maximum plasma concentration (Cmax).
Adverse Events | up to 9 weeks
  Safety and tolerability measure by number of subjects who experience adverse events
Safety Labs | up to 9 weeks
  Safety and tolerability measure by number of subjects who experience potential clinically significant changes in safety labs
ECGs | up to 9 weeks
  Safety and tolerability measure by number of subjects who experience potential clinically significant changes in ECGs
Vital Signs | up to 9 weeks
  Safety and tolerability measure by number of subjects who experience potential clinically significant changes in vital signs
Physical Examinations | up to 9 weeks
  Safety and tolerability measure by number of subjects who experience potential clinically significant changes in physical exams

CONTACTS AND LOCATIONS:
Overall Officials: Kirsteen Donaldson, FFPM,DM,FRCP, Study Director — Corcept Therapeutics
Locations (1):
- Celerion, Tempe, Arizona, United States